CLINICAL TRIAL: NCT04907123
Title: Systematic Escalation of diuREtics With Natriuresis in Heart Failure Patients: SERENA Trial
Acronym: SERENA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Simone Frea, MD, Cardiologist, A.O.U. Città della Salute e della Scienza - Molinette Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SERENA trial
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UNa+ Driven Intensive Therapy (Experimental): Ask patient to empty bladder. Start treatment (step 1). Re-evaluate patient every 6 hours; if therapeutic goal is not met, treat according to the following step.
  Therapeutic goal: Spot Urinary Sodium > 70 mEq/L AND mean diuresis > 1,5 ml/kg/h Step 1 Furosemide i.v. continuous infusion (2 times oral daily dose; minimum dose: 240 mg die) Step 2 Double furosemide i.v. continuous infusion (maximal dose: 720 mg die) Step 3 Add oral metolazone 5 mg b.i.d. Step 4 Add oral acetazolamide 250 mg b.i.d.
  Interventions: Other: Intensive sodiuria-guided diuretic treatment
- Standard Therapy (Active Comparator): Ask patient to empty bladder. Start treatment (step 1). Re-evaluate patient every 12 hours; if therapeutic goal is not met, treat according to the following step.
  Therapeutic goal: mean diuresis > 1,5 ml/kg/h Step 1 Furosemide i.v. continuous infusion (2 times oral daily dose; minimum dose: 240 mg die) Step 2 Double furosemide i.v. continuous infusion (maximal dose: 720 mg die) Step 3 Add oral metolazone 5 mg b.i.d. Step 4 Add oral acetazolamide 250 mg b.i.d.
  Interventions: Other: Standard diuretic treatment

INTERVENTIONS:
Other: Intensive sodiuria-guided diuretic treatment — Intensive stepwise diuretic treatment based on combined diuresis and urinary sodium assessment
  Arms: UNa+ Driven Intensive Therapy
Other: Standard diuretic treatment — Stepwise diuretic therapy based on diuresis assessment
  Arms: Standard Therapy

SUMMARY:
The present is a multicenter, prospective, randomized, open-label, blinded end-point trial aiming to investigate the clinical benefit of a stepwise, natriuresis-driven diuretic strategy versus standard diuretic treatment in patients with acute decompensated heart failure with reduced ejection fraction (HFrEF) and low early urinary sodium excretion. The study will focus on patients at increased risk of resistance to diuretic therapy. In particular, patients admitted to the emergency department and cardiac intensive care unit due to an on-chronic or de-novo acute decompensated HF episode with a predominantly "wet" profile and low early spot urinary sodium (UNa+) excretion will be considered. Spot natriuresis is a low-cost, non-demanding laboratory test in use to identify diuretic-resistant patients with an inherent poor prognosis. Whether the early identification of diuretic resistant patients and the consequent more aggressive treatment may lead to a better outcome has not been demonstrated by randomized studies. This trial aims to assess if an intensive stepwise diuretic approach guided by systematic urinary output assessment including natriuresis evaluation versus a standard diuretic strategy based on urinary output alone effectively leads to faster euvolemia achievement and better prognosis in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Admission for acute decompensate chronic heart failure or acute de novo heart failure
* Ejection Fraction <40%
* Severe signs and symptoms of congestion with modified wet score ≥ 12
* Spot urinary sodium excretion ≤ 70 mEq/L at 2 hours from first intravenous loop diuretic administration
* Systolic blood pressure ≥90 mmHg

Exclusion Criteria:

* Reversible etiology of acute heart failure (including acute coronary syndromes, myocarditis, acute pulmonary embolism, acute rhythm disorders, severe organic valve disease)
* Cardiogenic shock at admission or sign of hypoperfusion needing inotropic agents or mechanical circulatory support.
* eGFR lower than 15 ml/min/1.73m2 or dialysis
* Pregnancy or breastfeeding

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Evidence of significant reduction of congestion defined as absolute reduction of at least 1 point in wet score grading of congestion after 48 hours of treatment | 48 hours
  Assessment of WET score (Gheorghiade et al, EJHF 2010)

SECONDARY OUTCOMES:
Treatment failure, defined as persistent congestion (graded by wet score ≥12/20) after 24, 48 and 72 hours of diuretic treatment or need for renal replacement therapy. | 24,48 and 72 hours
Freedom from congestion at 48 hours, defined as jugular venous pressure of <8 cm, with no orthopnea and with trace peripheral edema or no edema | 48 hours
Worsening or persistent heart failure | 48 hours
  worsening heart failure symptoms or failure of the patient's condition to improve with treatment requiring the initiation of intravenous inotropic therapy and/or the implementation of mechanical circulatory or ventilatory support up until 48 hours
Composite endpoint of all-cause mortality, urgent LVAD implant or Heart Transplantation at 30 and 90 days. | 30 and 90 days
All-cause mortality | 30 and 90 days
Cardiac cause mortality | 30 and 90 days
  including myocardial infarction, irreversible heart failure, cardiogenic shock, fatal arrhythmic events
Rehospitalization for heart failure | 30 and 90 days
Worsening renal function | 48 hours
  absolute increase in serum creatinine > 0.3 mg/dl or > 1,5-fold from baseline at any time from randomization to 48 hours
Incidence of severe hypokalemia, severe hyponatremia or symptomatic electrolytes disorders during treatment protocol | 72 hours
  hypokalemia <3 mEq/L, severe hyponatremia <125 mEq/L
Severe symptomatic hypotension | 72 hours
  Systolic arterial pressure < 80 mmHg

OTHER OUTCOMES:
Time to oral switch of diuretic treatments | 90 days
  days
Time to discharge from hospital | 90 days
  days
Total Urinary output and urine output/40 mg furosemide | 24 and 48 hours
  ml/mg furosemide
Variation of body weight and body weight/40 mg furosemide | 24 and 48 hours
  kg/mg furosemide
Variation of NT-proBNP at 48 hours | 48 hours
Variation of wet score at 24 and 72 hours | 24 and 72 hours
Dyspnea severity variation at 24 and 48 hours assessed by dyspnea Visual Assessment Scale (VAS). | 24 and 48 hours
Fluid balance | 24, 48 and 72 hours
  In/out fluid balance
Time spent in Intensive Cardiac Intensive Care Unit | 90 days
  days

CONTACTS AND LOCATIONS:
Overall Officials: Simone Frea, MD, Principal Investigator — A.O.U. Città della Salute e della Scienza, Torino, Italia
Locations (1):
- A.O.U. Città della Salute e della Scienza di Torino, Torino, To, Italy